CLINICAL TRIAL: NCT06220942
Title: Tachycardia as an Indication for Prophylactic Phenylephrine Injection in Caesarean Section Under Spinal Anesthesia; an Observational Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, maha sadek El Derh, Assistant professor of Anesthesia, Ain Shams University
Other Study IDs: FMASUR338/2023
Record Dates: First submitted 2023-12-22; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Anesthesia
Keywords: Caesarean section , hypotension, spinal anesthesia, phenylephrine
MeSH Terms: conditions — Hypotension | interventions — Phenylephrine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Phenylephrine — Pregnant female presented for C.S. after receiving spinal anesthesia, recording the vital data, phenylephrine will be given in a dose of 50 µg IV immediately if the heart rate increases ≥ 20 % of baseline

SUMMARY:
The value of phenylephrine administration in response to tachycardia in preventing hypotension after spinal anesthesia in elective cesarean section.

DETAILED DESCRIPTION:
This observational study will take place at Ain Shams University Maternity hospitals, Cairo, Egypt. All patients will sign written informed consent before inclusion.

Sample size:

Using PASS 15 program for sample size calculation, setting confidence level at 95% and margin of error at 0.05, it is estimated that sample size of 80 women will be needed to detect an expected incidence rate of hypotension after phenylephrine administration of 30% "Hasanin et al., 2019"

Inclusion criteria:

ASA II pregnant female planned for elective C.S., aged between 18 -35 years old.

Exclusion criteria:

Emergency CS, Complicated CS (Severe bleeding, organ injury, uterine atony), ASA III, VI & patients with cardiovascular diseases For all pregnant females including whose in the study group, preoperative labs will be done including ( CBC, INR, Liver function & Kidney function) , oral and written informed consents will be taken from the patients with explanation of the spinal anesthesia and expected complications.

In OR wide pore IV access and preload started with crystalloids, full standard monitoring, spinal anesthesia will be performed by the expert anesthetist. The pregnant female will be in the sitting position and complete sterilization of her back, local anesthesia by 5 ml lidocaine 1% then the spinal needle (Pencil point 27 G) introduced between L4-5 and injection of (50 µg fentanyl + bupivacaine 0.5%) in total volume between 1.8 - 2.3 according to patient's height.

Then patient will lie supine with head elevated 30 degrees by a bellow and start recording the data just after spinal anesthesia.

Phenylephrine will be given in a dose of 50 µg IV immediately if the heart rate increases ≥ 20 % of baseline.

Then blood pressure & HR will be recorded after the administration of phenylephrine and every 5 minutes.

Any further doses given will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA II pregnant female planned for elective C.S., aged between 18 -35 years old.

Exclusion Criteria:

* Emergency CS, Complicated CS (Severe bleeding, organ injury, uterine atony), ASA III, VI patients with cardiovascular diseases

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant female at childbearing period
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Hypotension Avoidance of Hypotension Avoidance of Hypotension | all through the procedure (cesarean section)
  Measure number of hypotensive episodes that would occur after injection of prophylactic phenylephrine for caesarean section ,by spinal anesthesia

SECONDARY OUTCOMES:
Apgar score in neonates. Number of phenylephrine doses. Nausea & vomiting after spinal anesthesia. | all through the procedure (cesarean section)
  Measure Apgar score of neonate after delivery and compare the results with other neonate whose parturients that did not receive prophylactic phenylephrine

CONTACTS AND LOCATIONS:
Locations (1):
- maha sadek El Derh, Cairo, Heliopolis, Egypt

IPD SHARING:
Plan to Share IPD: Undecided